CLINICAL TRIAL: NCT02856412
Title: Improving Mind/Body Health and Functioning With Integrative Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1939-R
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Stress Disorders, Post-Traumatic; Exercise; Mindfulness
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Motor Activity | interventions — Salvage Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Veterans Group Exercise (Experimental): Exercise 3 times weekly (for 12 weeks), with each total workout lasting approximately 60 minutes. Integrative Exercise incorporates elements of strength training, flexibility, cardiovascular training, and controlled breathing exercises.
  Interventions: Other: Veterans Group Exercise (VGX)
- Illness Management and Recovery (Active Comparator): Attend 3 health education classes weekly (for 12 weeks), with each class lasting approximately 60 minutes. Illness Management and Recovery is an educational program focused on helping individuals more effectively manage their illnesses to pursue their personal recovery goals. The classes include the following topic areas which have been adapted for use in PTSD: recovery, practical facts about PTSD, stress-vulnerability, building social support, medications for PTSD, drug and alcohol use, reducing relapse, coping with stress, coping with persistent symptoms, getting needs met in the VA healthcare system, and living a healthy lifestyle.
  Interventions: Other: Illness Management and Recovery

INTERVENTIONS:
Other: Veterans Group Exercise (VGX) — Integrative Exercise incorporates elements of strength training, flexibility, cardiovascular training, and controlled breathing exercises.
  Other Names: VGX, Exercise Classes
  Arms: Veterans Group Exercise
Other: Illness Management and Recovery — Illness Management and Recovery is an educational program focused on helping individuals more effectively manage their illnesses to pursue their personal recovery goals. The classes include the following topic areas which have been adapted for use in PTSD: recovery, practical facts about PTSD, stress-vulnerability, building social support, medications for PTSD, drug and alcohol use, reducing relapse, coping with stress, coping with persistent symptoms, getting needs met in the VA healthcare system, and living a healthy lifestyle.
  Other Names: IMR, Health Education Classes, PTSD Recovery Classes
  Arms: Illness Management and Recovery

SUMMARY:
There is evidence demonstrating that aerobic exercise improves many symptoms of Posttraumatic Stress Disorder (PTSD) including; anxiety, depression, insomnia, and cognition. With the goal of using exercise as a rehabilitation therapy for Veterans with PTSD, a team of scientists and doctors developed a 12-week exercise program, combining aerobic and strength training with concentration training and mindful breathing techniques. The initial pilot study suggested that Integrative Exercise may improve overall quality of life, sleep quality, cardiovascular fitness, and PTSD symptoms. This new study will help determine the effectiveness of Integrative Exercise compared to health education classes. The overall goal is to determine if integrative exercise is an effective rehabilitation intervention for combat Veterans with PTSD.

DETAILED DESCRIPTION:
Despite the considerable efforts of the VA to improve awareness of mental health problems and access to care, many returning Veterans still report substantial barriers to seeking traditional mental health care. There is a large body of evidence demonstrating that aerobic exercise effectively improves many outcomes relevant to Posttraumatic Stress Disorder (PTSD) including; anxiety, depression, insomnia, cognition, and cardiovascular disease. In addition, there is a rapidly growing evidence base showing that aerobic exercise produces an increase in the growth of new neurons (e.g., neurogenesis) and increases the volume of the hippocampus which underscores the potential value of exercise for producing broad benefits to psychological health. Recognizing the promise that exercise might hold for attracting more Veterans into care and improving overall health in Veterans with PTSD, a team of investigators at the San Francisco Veterans Administration Medical Center (SFVAMC) with funding from the Department of Defense developed a treatment protocol and completed a pilot study of Integrative Exercise (Aerobic exercise and Breath Training 3 weekly sessions over 12 weeks) versus a waitlist control condition. Promising results from this trial have led us to the next step which is to conduct a definitive efficacy study of Integrative Exercise versus an active health education control condition: Illness Management and Recovery (IMR). The control condition will be matched on contact hours with treatment personnel. The goal of this revised proposal is to test if Integrative Exercise improves overall quality of life, PTSD symptoms, sleep quality, and measures of cardiovascular health in combat Veterans with chronic PTSD relative to the IMR condition. Another goal is to test if improvements in quality of life are predicted by improvements in cardiovascular fitness as measured by exercise capacity on treadmill testing. Finally, the proposal will test if Integrative Exercise versus IMR will produce greater improvements in additional health outcomes, including mood, subjective sleep quality, and PTSD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Veterans (Male and Female) between the ages of 18-75 who are physically able to participate in an exercise program
* Meet criteria for PTSD of at least 3 months duration, OR have some symptoms of PTSD with a current CAPS score of 23 or higher, as indexed by the Clinician Administered PTSD Scale for DSM-5 (CAPS-5)

Exclusion Criteria:

* History of any psychiatric disorder with active psychosis or mania in the past 5 years
* Meet criteria for severe drug or alcohol use disorder within the past 6 months as assessed by the Structured Clinical Interview for DSM-5
* Prominent suicidal or homicidal ideation
* Currently exposed to recurrent trauma or have been exposed to a traumatic event within the past 3 months
* Pregnant
* Have a clinically significant:

  * neurologic disorder
  * systemic illness affecting central nervous system (CNS) function
  * history of seizure disorder in the past 5 years
  * and/or physical disabilities making it impossible to use exercise equipment
* Acute coronary events (i.e., Myocardial Infarction) in the past 6 months
* Moderate to severe Traumatic Brain Injury (any history of head trauma associated with the onset of persistent cognitive complaints, neurological symptoms, or loss of consciousness > 30 minutes)
* Subjects who, in the opinion of the investigator, are otherwise unsuitable for a study of this type
* The investigators will not exclude patients with PTSD who are currently receiving individual or group therapy or patients who are currently taking antidepressant or anti-anxiety medication, but will apply the following criteria:

  * patients must have been in treatment for at least 2 months
  * meet symptomatic criteria for inclusion
  * do not have plans to discontinue treatment during the course of the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C. Neylan, MD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Neylan TC, Muratore LA, Williams CL, Schmitz M, Valdez CV, Maguen S, O'Donovan A, Kelley DP, Metzler TJ, Cohen BE, West AC, Phan JDV, Antonetti V, Mayzel O, Hlavin JA, Chesney MA, Mehling WE. Group integrated exercise versus recovery class for veterans with posttraumatic stress disorder: a randomized clinical trial. BMC Psychiatry. 2025 Feb 28;25(1):185. doi: 10.1186/s12888-025-06638-1. PMID 40021975

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Veterans Group Exercise | Illness Management and Recovery
Started | 41 | 43
Completed | 30 | 34
Not Completed | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Veterans Group Exercise | Illness Management and Recovery | Total
Number analyzed (Participants) | 41 | 43 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 43 | 84
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 30 | 28 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 5 | 14
  Not Hispanic or Latino | 27 | 32 | 59
  Unknown or Not Reported | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 9 | 21
  White | 18 | 26 | 44
  More than one race | 7 | 1 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 43 | 84

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale (CAPS) Score Comparison Between Subjects Randomized to Integrative Exercise Treatment vs. Illness Management and Recovery
Description: The CAPS-5 is a 20 item scale that provides both a dimensional and categorical measure of PTSD. The CAPS-5 items are rated with a single severity score, ranging from 0-80 with higher scores indicating worse severity, that incorporates both frequency and intensity PTSD-related symptoms. In addition to assessing the 20 DSM-5 PTSD symptoms, questions target the onset and duration of symptoms, subjective distress, impact of symptoms on social and occupational functioning, improvement in symptoms since a previous CAPS administration, overall response validity, overall PTSD severity, and specifications for the dissociative subtype (depersonalization and derealization).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Veterans Group Exercise | Illness Management and Recovery
Number analyzed (Participants) | 41 | 43
units on a scale | 24.4 (11.1) | 22.0 (11.3)

2. Primary Outcome: The World Health Organization Quality of Life (WHOQOL-BREF) Score Comparison Between Subjects Randomized to Integrative Exercise Treatment vs. Monitor Only
Description: The WHOQOL-BREF instrument comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment. The WHOQOL-BREF is a shorter version of the original WHOQOL-100 instrument and is more convenient for use in large research studies or clinical trials. The Psychological Domain, the investigators' primary outcome, is derived from 6 items which index body image, negative & positive feelings, self-esteem, spirituality, and cognition. Each of the 6 items have 5 response options with higher scores indicating higher psychological health. The mean score of items within each domain is used to calculate the domain score. The domain score is then linearly transformed to scale of 0-100 to enable comparisons between other domains composed of unequal numbers of items. (Skevington et al. Quality of Life Research 13: 299-310, 2004.)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Veterans Group Exercise | Illness Management and Recovery
Number analyzed (Participants) | 41 | 43
units on a scale | 41.5 (19.4) | 45.2 (16.8)

3. Secondary Outcome: Five Facet Mindfulness Questionnaire (FFMQ)- Observing
Description: The FFMQ is a 39-item questionnaire derived from a factor analysis of other mindfulness questionnaires. It assesses five facets of mindfulness: observing, describing, acting with awareness, non-judging and non-reactivity to inner experience which represent elements of mindfulness as it is currently conceptualized. Items are rated on a Likert scale ranging from 1 (never or very rarely true) to 5 (very often or always true). Scale range is 39-195 with higher scores indicating higher mindfulness. Score ranges for five facets are: observing (8-40; describing (8-40), acting with awareness (8-40), non-judging (8-40), and nonreactivity to inner experience (7-35).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Veterans Group Exercise | Illness Management and Recovery
Number analyzed (Participants) | 41 | 43
score on a scale | 22.2 (11.4) | 26.4 (7.1)

4. Secondary Outcome: Godin Leisure-Time Exercise Questionnaire
Description: The Godin Leisure-Time Exercise Questionnaire is a validated brief inventory assessing sedentary, work, recreational, and aerobic activity in a typical week. The overall score is between zero and 119, and higher GLTEQ scores demonstrate more physical activity.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Veterans Group Exercise | Illness Management and Recovery
Number analyzed (Participants) | 41 | 43
score on a scale | 44.2 (40.2) | 43.8 (36.0)

5. Secondary Outcome: PTSD Checklist for DSM-5 (PCL-5)
Description: The PCL-5 is a validated self-report rating scale for assessing PTSD symptoms. It consists of 20 items that correspond to the DSM-5 symptoms of PTSD. The range is 0-80 with higher scores indicating worse severity.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Veterans Group Exercise | Illness Management and Recovery
Number analyzed (Participants) | 41 | 43
score on a scale | 36.3 (17.5) | 39.9 (15.7)

6. Secondary Outcome: Symptom Check-List-90-Revised (SCL-90-R)
Description: The SCL-90-R is a standard self-report measure of general psychopathology. Each item on the SCL-90-R is graded on a five-point scale from 0 (not at all) to 4 (extremely).The Global Severity Index (GSI) is the average score for all the items and ranges from 0-4 with higher scores indexes greater psychopathology.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Veterans Group Exercise | Illness Management and Recovery
Number analyzed (Participants) | 41 | 43
score on a scale | 1.14 (0.68) | 1.13 (0.57)

7. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: This self-report measure provides a subjective assessment of sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances (including nightmares), use of sedative-hypnotics, and daytime energy. The PSQI global score range is 0-21 with higher scores indicating worse sleep quality.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Veterans Group Exercise | Illness Management and Recovery
Number analyzed (Participants) | 41 | 43
score on a scale | 11.4 (5.2) | 10.7 (4.2)

8. Secondary Outcome: Insomnia Severity Index (ISI)
Description: The ISI is a self-report measure that is a more specific index of perceived insomnia severity, as compared to the widely used PSQI measure which captures sleep disturbances of all types. The ISI uses a 5-point Likert scale to rate the severity of insomnia symptoms. The total score ranges from 0-28 with higher scores indicating worse insomnia severity.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Veterans Group Exercise | Illness Management and Recovery
Number analyzed (Participants) | 41 | 43
score on a scale | 13.6 (6.8) | 13.2 (5.4)

ADVERSE EVENTS:
Time Frame: AEs, SAEs, and UAPs were collected from the time of study entry until the end of study participation which ranged from 12-24 weeks.
Arm/Group | Veterans Group Exercise | Illness Management and Recovery
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/43
Other Adverse Events (participants affected / at risk) | 0/41 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/12/NCT02856412/Prot_SAP_000.pdf